CLINICAL TRIAL: NCT02595840
Title: Biomarker Study Accompanying the AIO-TRK-0114 Study (MARBLE)
Acronym: Trans-MARBLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Martin Schuler, Prof. Dr. med., Director, Department of Medical Oncology, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT-Nr. 2014-001983-36
Record Dates: First submitted 2015-10-23; First posted 2015-11-04 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Non-small-cell Lung Cancer With Somatic EGFR Mutations
MeSH Terms: interventions — Afatinib; Pemetrexed

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Afatinib (Experimental): Afatinib 40 mg/d (30, or 20 mg/d in case of dose reduction during 1st line treatment)
  Interventions: Drug: Afatinib
- Arm B: Pemetrexed (Experimental): Pemetrexed 500 mg/m2 (375 mg/m² in case of dose reduction during induction therapy) i.v. on d1 of each 21-day cycle
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Afatinib
  Arms: Arm A: Afatinib
Drug: Pemetrexed
  Arms: Arm B: Pemetrexed

SUMMARY:
To compare the efficacy of afatinib maintenance with pemetrexed maintenance following induction therapy with platinum/ pemetrexed in patients with metastatic EGFR mutated non-small-cell lung cancer progressing after first-line treatment with afatinib as first tyrosine kinase inhibitor with respect to progression-free survival

DETAILED DESCRIPTION:
Patients who have progressed after first-line treatment with afatinib as first tyrosine kinase inhibitor (TKI) will be screened while they are receiving second-line (induction) treatment consisting of cisplatin / carboplatin plus pemetrexed given in 21-day cycles. Patients who do not progress (i.e. complete or partial response, or stable disease - CR, PR or SD) after completion of at least three and not more than four chemotherapy cycles will be randomized (1:1 ratio) to receive maintenance therapy with either afatinib (40 mg/d or last tolerated dose during first-line treatment with afatinib as first TKI) or pemetrexed (500 mg/m2 or 375 mg/m2 if dose reduction was required every 21 days) until disease progression or treatment discontinuation because of patient decision or toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in the AIO-TRK-0114 (MARBLE) study (EudraCT-No. 2014-001983-36)
2. Written informed consent

Exclusion Criteria:

1. Patients who do not meet the inclusion criterial of the AIO-TRK-0114 (MARBLE) study (EudraCT-No. 2014-001983-36)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival in relation to exploratory biomarkers | until progression

SECONDARY OUTCOMES:
Overall Survival in relation to exploratory biomarkers | continuous assessment
  Overall survival
Objective response rate | Assessed every 6 weeks for 24 weeks, then every 9 weeks
  Objective response rate, clinical benefit rate (RECIST 1.1)